CLINICAL TRIAL: NCT05954468
Title: Psycho-social Impact of Anti-NMDAR Encephalitis
Acronym: SAPIENCE
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL21_0628
Record Dates: First submitted 2023-07-13; First posted 2023-07-20 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: NMDAR Antibody-associated Auto-immune Encephalitis
Keywords: auto-immune encephalitis; NMDA receptor encephalitis; Health-related quality of life; psyco-social impact; cognitive consequence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: standardized and validated surveys — To evaluate the cognitive and psycho-social long term impact of a NMDAR encephalitis, we will collect the data using specific interview assessments such as the PROMS (Patient-reported Outcome Measures Information System) and PREMS (Patient-reported experiences measures) as well as we will check the cognitive performance in order to combine the expertise from clinical neurology, social & health psychology

SUMMARY:
NMDA receptor encephalitis is a rare neurological autoimmune disease with severe neuropsychiatric symptoms, but a typically good functional neurological outcome. The majority of patients experience long-term cognitive, psychological and social impairments that have significant consequences for their well-being and quality of life. However, as the disease was only recently discovered (Dalmau and al. Annals of neurology, 2007), this psycho-social impact has not been studied systematically and the resulting consequences for patients are not adequately appreciated.

The proposed study aims at characterizing the cognitive and psycho-social long-term consequences of this rare disease. Our main hypothesis is that NMDAR encephalitis has a persistent and clinically relevant impact on the patients' long-term cognitive, psychological and social well-being. Furthermore, we hypothesize that longterm subjective outcomes depend on both internal and external factors, such as acute disease course, access to post-acute care, caregiver support, personal coping strategies, or access to health education resources and peer group support.

ELIGIBILITY:
Inclusion Criteria:

* Patients with anti-NMDAR encephalitis
* Year ≥ 18 ans
* Patients affiliated to the social security scheme

Exclusion Criteria:

* Patients with no anti-NMDAR encephalitis
* Minor patient
* Patient under guardianship or curatorship
* Patient with preexisting neurological symptoms

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study involves patients with autoimmune encephalitis with anti-NMDAR antibodies.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2023-10-09 (Actual); Primary Completion 2024-09-04 (Actual); Study Completion 2024-09-04 (Actual)

PRIMARY OUTCOMES:
Cognitive and psycho-social analyses of patients with NMDAR encephalitis. | At study completion in an average of 12 months
  The analyze will focus on the post-acute phase of the disease.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre de référence des syndromes neurologiques paranéoplasiques et encéphalites auto-immunes, Hôpital neurologique Pierre Wertheimer, Bron, Bron, France

IPD SHARING:
Plan to Share IPD: No